CLINICAL TRIAL: NCT02230761
Title: A Phase 2, Randomized, Double-masked, Placebo-controlled Study of XOPH5 Ointment for Reduction of Lower Lid Steatoblepharon
Brief Title: Phase 2 Study of XAF5 (XOPH5) Ointment for Reduction of Excess Eyelid Fat (Steatoblepharon)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XOPH5-OINT-2
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2015-12

CONDITIONS: Lower Eyelid Steatoblepharon (Excess Eyelid Fat)
Keywords: steatoblepharon; blepharoptosis; dermatochalasis; blepharoplasty; periorbital; orbital; eyelid; eyebags; eye bags
MeSH Terms: conditions — Blepharoptosis; Cutis Laxa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- XOPH5 Ointment (Experimental): XOPH5 Ointment is the investigational drug to be studied.
  Interventions: Drug: XOPH5 Ointment
- Placebo Ointment (Placebo Comparator): Placebo is an ointment that matches XOPH5 Ointment but lacks the active ingredient.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XOPH5 Ointment
  Arms: XOPH5 Ointment
Drug: Placebo
  Arms: Placebo Ointment

SUMMARY:
This study will test whether XAF5 (XOPH5) ointment, applied once daily to the lower eyelids for 10 weeks, reduces the prominence of lower eyelid fat in adults with moderate to severe steatoblepharon (excess eyelid fat).

ELIGIBILITY:
Inclusion Criteria (abbreviated):

* Moderate to severe lower eyelid steatoblepharon (LESS score of 2-4 bilaterally)
* Men and women 40-70 years old
* Healthy facial skin
* Must understand and provide informed consent

Exclusion Criteria (abbreviated):

* Best corrected visual acuity worse than 20/40 in either eye
* Regular use of ophthalmic medication in either eye
* Planned use of contact lenses during the study
* Any history of lower eyelid surgery

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S. Singer, MD, PhD, Study Chair — Topokine Therapeutics, Inc.
Locations (1):
- Topokine Therapeutics Clinical Study Centers, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- XOPH5 Ointment: XOPH5 Ointment is the investigational drug to be studied.
  XOPH5 Ointment
- Placebo Ointment: Placebo is an ointment that matches XOPH5 Ointment but lacks the active ingredient.
  Placebo
Period: Overall Study
Arm/Group | XOPH5 Ointment | Placebo Ointment
Started | 60 | 30
Completed | 60 | 29
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XOPH5 Ointment | Placebo Ointment | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.2 (7.4) | 55.1 (7.5) | 54.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 17 | 57
  Male | 20 | 13 | 33

OUTCOME MEASURES:

1. Primary Outcome: Lower Eyelid Steatoblepharon Severity (LESS) Score--Clinician-Reported
Description: Photonumeric scale, range 0-4, 0 is absence of steatoblepharon, 4 is very severe steatoblepharon.
Time Frame: 11 weeks
Population: intention-to-treat
Measure: Number; unit: participants
Arm/Group | XOPH5 Ointment | Placebo Ointment
Number analyzed (Participants) | 60 | 30
participants | 27 | 6
Statistical Analysis 1: Comparison: XOPH5 Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.020, Chi-squared

2. Other Pre Specified Outcome: Patient Satisfaction Scale 1 (PSS1)
Description: Change from Baseline to Week 11 in PSS1 score. PSS1 scale items use an ordinal scale with range 0-10, where 0 is the least favorable and 10 is the most favorable. The composite score is the sum of 6 items and has a possible response range of 0 to 60.
Time Frame: 0-11 weeks
Population: intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XOPH5 Ointment | Placebo Ointment
Number analyzed (Participants) | 60 | 30
units on a scale | 17.9 (14.4) | 7.3 (13.0)
Statistical Analysis 1: Comparison: XOPH5 Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.001, t-test, 2 sided

3. Other Pre Specified Outcome: Patient Satisfaction Scale 2 (PSS2)
Description: Composite score on PSS2 scale. PSS2 is an ordinal scale with range 1-7, where 1 is least favorable and 7 is most favorable. The composite score is the sum of 3 items and has a possible response range of 3 to 21.
Time Frame: 11 weeks
Population: intention-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | XOPH5 Ointment | Placebo Ointment
Number analyzed (Participants) | 60 | 30
units on a scale | 16.3 (3.3) | 14.0 (3.0)
Statistical Analysis 1: Comparison: XOPH5 Ointment vs Placebo Ointment; Test type: Superiority or Other; p = 0.002, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | XOPH5 Ointment | Placebo Ointment
Serious Adverse Events (participants affected / at risk) | 0/60 | 1/30
Other Adverse Events (participants affected / at risk) | 11/60 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XOPH5 Ointment (N=60) | Placebo Ointment (N=30)
Guillan-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XOPH5 Ointment (N=60) | Placebo Ointment (N=30)
Hyperemia eyelid (mild, transient) (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Increase in vellus hair (mild) (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less